CLINICAL TRIAL: NCT07101471
Title: A Prospective and Observational Study for Safety and Effectiveness Evaluation of Rhofanib® (Tofacitinib) in Patients With Alopecia.
Brief Title: Rhofanib® (Tofacitinib) Safety and Effectiveness Evaluation
Status: Completed | Type: Observational
Sponsor: NanoAlvand (Industry)
Responsible Party: Sponsor
Other Study IDs: RHO.NA.SD.IV.99
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Alopecia Totalis/Universalis; Alopecia Areata(AA)
Keywords: tofacitinib; Alopecia Areata; Severity of Alopecia Tool score; Alopecia Universalis; Alopecia Totalis
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants received Rhofanib® (Tofacitinib)
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib with a suggested dose of 5 mg twice daily with or without adjuvant prednisolone.

SUMMARY:
The goal of this observational study is to evaluate safety of Rhofanib® (Tofacitinib) in male or female participants with the age of 18 years or older having clinical diagnosis of Alopecia. The main questions are aim to answer:

1. Is Rhofanib® (Tofacitinib) safe in Alopecia?
2. Is Rhofanib® (Tofacitinib) work to treat Alopecia?

In this study, there is no comparison group. Participants received Rhofanib® (Tofacitinib) with or without adjuvant prednisolone.

DETAILED DESCRIPTION:
This study is a phase IV, post-marketing, observational, cohort study for the safety and effectiveness evaluation of Rhofanib® (Tofacitinib) use in Iranian participants with alopecia with at least 40% scalp hair loss, alopecia totalis, or alopecia universalis.

Researchers and investigators gathered data in booklets. Exposure to Rhofanib® (Tofacitinib) in this study was defined as administration of Rhofanib® (Tofacitinib) with a suggested dose of 5 mg twice daily with or without adjuvant prednisolone.

The primary objective of this study was safety assessment, including the incidence of the most common adverse events (AEs), serious adverse events, and death during the study period.

The secondary objective is the effectiveness of Rhofanib® (Tofacitinib) by assessment of the Severity of Alopecia Tool (SALT) score, disease relapse (Patchy or complete scalp hair loss), eyebrow and eyelash status affected by alopecia, and also participants' quality of life-based on Dermatology life quality index (DLQI) during the study period.

This study was a single arm and the sample size of this study was 353 participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with the age of 18 years or older
* Clinical diagnosis of alopecia areata with at least 40% scalp hair loss, alopecia totalis, or alopecia universalis who are prescribed Rhofanib®
* Stable or worsening disease for at least 6 months
* Patients who have given written authorization to use their personal health data for the purpose of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Safety assessment | Study period ( Up to 6 months)
  Safety assessment, including the incidence of AEs. All AEs are classified based on the Medical Dictionary for Regulatory Activities (MedDRA Desktop Browser 4.0 Beta) terms as System Organ Class (SOC) and Preferred Term (PT). All the reported events are graded according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). Moreover, seriousness of AEs is assessed according to International Council for Harmonisation (ICH-E2B) guidelines. The causality relation is assessed based on the World Health Organization (WHO) criteria.

SECONDARY OUTCOMES:
The percentage of change from baseline in the Severity of Alopecia Tool (SALT) Score | Study period (up to 6 months)
  Severity of Alopecia Tool (SALT) Score is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss).
The frequency of relapse disease (Patchy or complete scalp hair loss). | Study period (up to 6 months)
The frequency and proportion of participants achieved greater or equivalent to one grade improvement in eyelash/ eyebrow scores | Study period (up to 6 months)
  It is a 4-point scale that is used to assess the severity of eyebrow and eyelash hair loss in Alopecia, with the scale ranging from 0 to 3. The score of 0 equals to worth case, and the score of 3 indicates normal.
Change in Dermatology Life Quality Index Total Score (DLQI) | Study period (up to 6 months)
  Dermatology Life Quality Index Total Score (DLQI) is a questionnaire that ranges from 0 to 30. Higher scores indicate a greater negative impact on quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Orchid Pharmed, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
Data produced in the present study are available upon reasonable request from the investigators.

REFERENCES:
- [Background] Wohltmann WE. JAAD Game Changers: Tofacitinib for the treatment of severe alopecia areata and variants: A study of 90 patients. J Am Acad Dermatol. 2024 Nov;91(5):825. doi: 10.1016/j.jaad.2024.05.064. Epub 2024 May 31. No abstract available. PMID 38823686
- [Background] Liu LY, King BA. Tofacitinib for the Treatment of Severe Alopecia Areata in Adults and Adolescents. J Investig Dermatol Symp Proc. 2018 Jan;19(1):S18-S20. doi: 10.1016/j.jisp.2017.10.003. PMID 29273099
- [Background] Liu LY, Craiglow BG, Dai F, King BA. Tofacitinib for the treatment of severe alopecia areata and variants: A study of 90 patients. J Am Acad Dermatol. 2017 Jan;76(1):22-28. doi: 10.1016/j.jaad.2016.09.007. Epub 2016 Nov 2. PMID 27816293